CLINICAL TRIAL: NCT03213613
Title: Double-Blind Randomized Controlled Trial for the Evaluation of a Novel Adaptive Attention Training in Healthy Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Alliance for Decision Education (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: P0505751
Record Dates: First submitted 2017-07-07; First posted 2017-07-11 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Healthy Adolescents
Keywords: Teen health; Teen development; Adolescent development; Memory; Attention; Reward processing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Adaptive Attention Training (Experimental): The training group will engage in 15 hours of at-home training on a novel iPad-based adaptive attention training program ('Engage'). Individuals will complete thirty 30-minute sessions over six weeks. Training compliance and performance data (accuracies and reaction times) will be continuously monitored remotely and analyzed over secure online servers to ensure that participants are completing training as scheduled and to deal with any unexpected road-blocks in training.
  Interventions: Behavioral: Adaptive Attention Training
- Active Control (Placebo Comparator): The active control group will engage in 15 hours of at-home training on an iPad game ('Boing'). Individuals will complete game play for the same number of hours as the training group to control for the effects of computer exposure and interaction, contact with research personnel, and monetary rewards. Compliance will be monitored similarly to the adaptive attention training group.
  Interventions: Behavioral: Active Control
- Low-dose Adaptive Attention Training (Placebo Comparator): The low-dose training group will engage in 1 hour of at-home training on 'Engage'. Individuals will complete two 30-minute sessions at the beginning and middle of a six-week period. Compliance will be monitored similarly to the adaptive attention training group.
  Interventions: Behavioral: Low-dose Adaptive Attention Training

INTERVENTIONS:
Behavioral: Adaptive Attention Training — The training is comprised of a time-based titration of rich audiovisual and sparse audio interactive environments. Training progressively transitions the participants from an immersive and rapid reward setting to a less immersive, sensory impoverished, and slower reward setting. Further, the participants' actions require delayed gratification decisions to accomplish play in the sparse setting, building fronto-parietal control through sustained attention and suppression of ventral-striatal reward impulses.
  Arms: Adaptive Attention Training
Behavioral: Active Control — Participants in the expectancy-matched active control group will play a visuo-spatial iPad game, in which players use their finger to move an object to different successive square platforms. Expectancy matching to the adaptive attention training was pre-confirmed in 121 participants (18-20 years of age), using targeted surveys on MTurk about their expectations of either training exposure on our specific outcome measures. To balance expectations of potential benefits, this group will receive identical recruitment and experimental instructions as the adaptive attention training group.
  Arms: Active Control
Behavioral: Low-dose Adaptive Attention Training — Participants in the low-dose training group will play a reduced number of sessions as the Adaptive Attention Training group. Specifically, they will train for two 30-minute sessions at the start and middle of a six-week period. To balance expectations of potential benefits, this group will receive identical recruitment and experimental instructions as the adaptive attention training group.
  Arms: Low-dose Adaptive Attention Training

SUMMARY:
This project will evaluate the neuro-cognitive outcomes of a novel, adaptive attention training in a healthy adolescent population.

DETAILED DESCRIPTION:
Aspects of cognitive control, such as attention and working memory, are critical for successful goal-directed behavior. Importantly, variability in cognitive control abilities can influence real-world functioning, such as scholastic success in children and adolescents. The primary goal of this project is to examine the outcomes of a novel, adaptive attention training that primarily targets aspects of sustained attention and secondarily targets delayed gratification in adolescents. As such, the investigators will validate the feasibility and efficacy of this novel training in a randomized controlled trial (RCT) study. Specifically, healthy adolescents (age 12-16 years old) will be recruited for a longitudinal experiment in which they are randomly assigned to the adaptive attention training group ('Engage') or one of two expectancy-matched control groups. Depending on the assigned group, participants will complete 1 hour (low-dose control group) or 15 hours ('Engage' and active control groups) of training as well as pre-, post- and follow-up assessments of cognitive, neural, and behavioral measures. We hypothesize that completion of 'Engage' training will result in enhancement of fronto-parietal control functions that underlie sustained attention and suppression of ventral-striatal reward impulses, ultimately improving these abilities in a healthy adolescent population.

ELIGIBILITY:
Inclusion Criteria:

* Healthy right-handed children, age 12-16 years old
* No ADHD status (verified with the Vanderbilt ADHD Parent form)
* Willing and able to undergo MRI and EEG procedures

Exclusion Criteria:

* Current psychotropic medications
* Current diagnosis of any axis I psychiatric disorder
* History of seizure disorder or seizure episodes over the last 2 years
* Motor/perceptual handicap that prevents computer use

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2022-12-13 (Actual); Study Completion 2022-12-13 (Actual)

PRIMARY OUTCOMES:
Test of Variables of Attention (TOVA), visual form, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.

SECONDARY OUTCOMES:
Delay Discounting task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.

OTHER OUTCOMES:
Filter task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of visual working memory with distraction
Attend Ignore Distractor (AID) task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of visual working memory with distraction during memory delay
Adaptive Cognitive Evaluation (ACE) neuropsychological battery, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For global assessment of cognitive control
EEG-based neural processing of stimuli in Test of Variables of Attention (TOVA), visual form, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of neural processing underlying sustained attention
fMRI-based blood oxygen level dependent (BOLD) signal processing during Delay Discounting task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of neural processing underlying delay discounting
EEG-based neural processing of stimuli in Filter task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of neural processing underlying visual working memory with distraction
EEG-based neural processing of stimuli in Attend Ignore Distractor (AID) task, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of neural processing underlying visual working memory, with distraction during memory delay
Resting-state functional connectivity (functional MRI and EEG), change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For neural assessment of intrinsic functional connections between brain regions
Structural connectivity (diffusion tensor imaging, DTI), change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For neural assessment of structural (white matter) connections between brain regions
Mindful Attention Awareness Scale (MAAS), change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For behavioral assessment of mindful attention awareness
Warwick-Edinburgh Mental Wellbeing-Scale, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For behavioral assessment of mental wellbeing
Torrance Tests of Creative Thinking, change from baseline | Change from baseline at completion of practice on assigned intervention.
  For assessment of visual creativity
Child Self-Control Rating Scale (parent and teacher ratings), change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For behavioral assessment of self-control
SEA battery, change from baseline | Change from baseline at completion of practice on assigned intervention and at 6 months follow-up post-intervention.
  For assessment of math and reading skills

CONTACTS AND LOCATIONS:
Overall Officials: Courtney Gallen, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- UCSF Neuroscape, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No